CLINICAL TRIAL: NCT03877965
Title: Pharmacokinetics and Safety Profile of Digoxin in Infants With Single Ventricle Congenital Heart Disease
Acronym: DGX01
Status: Completed | Type: Observational
Sponsor: Christoph P Hornik, MD MPH (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Christoph P Hornik, MD MPH, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00102130; NICHD-2018-DGX01 (Other: Duke); HHSN27500002 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Digoxin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected to assess pharmacokinetic and biomarker levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with single ventricle congenital heart disease: Receiving digoxin per standard of care during the interstage period
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — Drug administered per standard of care, with a dosing regimen within the labeled dose range of 7.5-20 mcg/kg/day divided in 2 or 3 equal doses

SUMMARY:
This is a prospective, multi-center, open-label, PK and safety profile study of enteral digoxin in children <6 months old at time of enrollment, post-surgical or hybrid stage 1 palliation, but prior to surgical stage 2 palliation.

DETAILED DESCRIPTION:
The Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) funded this protocol titled "Pharmacokinetics and Safety Profile of Digoxin in Infants with Single Ventricle Congenital Heart Disease", protocol number NICHD-2018-DGX01. The Investigational New Drug (IND) Sponsor and Principal Investigator for this protocol is Christopher P. Hornik, MD, MPH. The Contracting Officer's Technical Representative (COTR) to represent the Government for this task order is Perdita Taylor-Zapata. The Duke IRB number for this study is Pro00102130. This study employs a central IRB, the WIRB-Copernicus Group (WCG). The c-IRB (WCG) study number is 20190888 / NICHD-2018-DGX01.

This is a prospective, multicenter Phase 1 study with a primary objective to characterize the pharmacokinetics of enteral digoxin in infants with single ventricle congenital heart disease. The secondary objective is to determine the safety profile of enteral digoxin in infants with single ventricle congenital heart disease. Digoxin is used for the treatment of heart failure in pediatric patients and acts by controlling numerous functions of the cardiovascular system. Digoxin use in single ventricle congenital heart disease may decrease interstage mortality.

The study will be conducted in approximately 48 subjects at approximately 13 investigational centers. The proposed duration of the study is approximately 196 (±) days.

Please see the protocol and synopsis for more information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of single ventricle congenital heart disease
* Status post-surgical or hybrid stage 1 palliation but prior to surgical stage 2 palliation
* Age ≤ 30 days of life at time of stage 1 palliation
* Age < 6 months at time of enrollment
* Require treatment with enteral digoxin per their treating medical provider if their planned maintenance treatment dosing regimen is within the labeled dose range of 7.5 - 20 mcg/kg/day divided in 2 or 3 equal doses
* Informed consent from parent(s) or legal guardian(s)

Exclusion Criteria:

* Serum creatinine > 2 mg/dL at enrollment
* Diagnosis of second degree or higher atrioventricular conduction block at enrollment
* Diagnosis of clinically significant sinus bradycardia requiring intervention at enrollment
* Known hypersensitivity to digoxin or other forms of digitalis
* Extracorporeal life support (i.e., ECMO, dialysis, ventricular assist device) at enrollment
* Received digoxin prior to enrollment
* Received or anticipated to receive a loading dose of digoxin.
* Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study

Max Age: 6 Months | Sex: All
Age Groups: Child
Study Population: Up to 48 infants diagnosed with single ventricle congenital heart disease, receiving digoxin per standard of care during the interstage period
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of digoxin | Approximately 7 months
  The primary outcome measures are plasma concentrations of digoxin measured using a validated bioanalytical assay at a central laboratory.

SECONDARY OUTCOMES:
Number of adverse events related to study procedures and serious, unexpected, suspected adverse reactions related to digoxin | Approximately 7 months
  1. Adverse events (AEs) related to the study procedures (blood draws and outcome assessments), and serious, unexpected, suspected adverse reactions (SUSARs) related to digoxin will be captured.
Tachyarrthmias | Approximately 7 months
  Event of special interest will be captured (number of tachyarrythmias)
Number of participants with second and third degree atrioventricular conduction block | Approximately 7 months
Number of participants with sinus bradycardia | Approximately 7 months
  Number of participants with sinus bradycardia
Number of participants with need for temporary or permanent pacing | Approximately 7 months
  Number of participants with need for temporary or permanent pacing
Frequency of death | Approximately 7 months
  Frequency of death
PR interval | Approximately 7 months
  Derived from electrocardiograms and their reports performed per standard of care
QRS duration | Approximately 7 months
  Derived from electrocardiograms and their reports performed per standard of care
QT interval | Approximately 7 months
  Derived from electrocardiograms and their reports performed per standard of care
Corrected QT interval using Bazett's formula | Approximately 7 months
  Derived from electrocardiograms and their reports performed per standard of care

OTHER OUTCOMES:
Plasma concentration of NT-proBNP | Approximately 7 months
Plasma concentration of MR-proANP | Approximately 7 months
Right ventricular or left ventricular end diastolic volume | Approximately 7 months
Right ventricular or left ventricular end systolic volume | Approximately 7 months
Right ventricular or left ventricular ejection fraction | Approximately 7 months
Right ventricular or left ventricular shortening fraction | Approximately 7 months
Right ventricular or left ventricular end diastolic dimension | Approximately 7 months
Right ventricular or left ventricular end systolic dimension | Approximately 7 months
Right ventricular or left ventricular fractional area change | Approximately 7 months
Degree of atrioventricular valve regurgitation | Approximately 7 months
Qualitative right ventricular or left ventricular function assessment | Approximately 7 months
Cardiac output | Approximately 7 months
  As measured by cardiac catheterization
Pulmonary to systemic blood flow ratio | Approximately 7 months
  As measured by cardiac catheterization
Pulmonary vascular resistance | Approximately 7 months
  As measured by cardiac catheterization
Mean pulmonary artery pressure | Approximately 7 months
  As measured by cardiac catheterization
Right ventricular or left ventricular end diastolic pressure | Approximately 7 months
  As measured by cardiac catheterization
Right ventricular or left ventricular end systolic pressure | Approximately 7 months
  As measured by cardiac catheterization
Right and left pulmonary artery size | Approximately 7 months
  As measured by cardiac catheterization
Pressure gradients across the aortic arch | Approximately 7 months
  As measured by cardiac catheterization
Incidence of unplanned surgical intervention | Approximately 7 months
  Including cannulation for mechanical circulatory support
Incidence of listing for heart transplant | Approximately 7 months
Incidence of receiving heart transplant | Approximately 7 months
Hospital length of stay after S1P | Approximately 7 months
Number of days on mechanical ventilation after S1P | Approximately 7 months
Number of hospital readmissions from S1P discharge to S2p | Approximately 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, MD, Principal Investigator — Duke University
Locations (11):
- United States (11):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Rady Childrens Hospital and Health Center, San Diego, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Nicklaus Children's Hospital, Miami, Florida
  - St. Louis Children's Hospital, St Louis, Missouri
  - Morgan Stanley Children's Hospital of New York Presbyterian, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No